CLINICAL TRIAL: NCT03933657
Title: Prospective Study on the Clinical Effectiveness, Safety, Cost Benefits, and Outcomes of the SoundBite™ Crossing System in Complex Peripheral CTOs - The PROSPECTOR II Study
Brief Title: Prospective Study of the SoundBite™ Crossing System in Complex Peripheral CTOs
Acronym: PROSPECTORII
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Replaced by CaTO-PAD/BTK Study
Sponsor: SoundBite Medical Solutions, Inc. (Industry)
Collaborators: ethica Clinical Research Inc. (Industry); Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT-PER-2019-01
Record Dates: First submitted 2019-04-24; First posted 2019-05-01 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Peripheral Arterial Occlusive Disease; Chronic Total Occlusion of Artery of the Extremities
Keywords: Chronic Total Occlusion; CTO; Crossing Device; Peripheral; SoundBite Crossing System
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Intervention Model Description: The population includes subjects with documented symptomatic peripheral CTOs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SoundBite™ Crossing System - Peripheral (Experimental): SoundBite™ Crossing System-Peripheral is indicated to facilitate the intraluminal placement of conventional guidewires or treatment devices beyond peripheral artery chronic total occlusions via atherectomy.
  Interventions: Device: SoundBite™ Crossing System - Peripheral

INTERVENTIONS:
Device: SoundBite™ Crossing System - Peripheral — SoundBite™ Crossing System consisting of the SoundBite™ Console and SoundBite™ Active Wire 18. The Investigator may use the SoundBite™ Active Wire during the procedure to cross the proximal aspect and/or to cross multiple lesions.

SUMMARY:
This study aims at assessing additional performance characteristics of the SoundBite™ Crossing System with regards to the luminal passage of complex Chronic Total Occlusions (CTO) by evaluating clinically relevant efficacy, safety, cost benefit and treatment pathway endpoints.

DETAILED DESCRIPTION:
This multinational study will be based on observational cases with descriptive statistics to collect data on safety and efficacy based on clinical use of the SoundBite™ Crossing System.

This study will include a cost benefit analysis that will focus on wire and other Percutaneous Transluminal Angioplasty (PTA) device usage during the procedure. The cost benefit will be compared to the sites data on their average costs for CTO crossing cases.

The planned treatment pathway elected prior to procedure will be compared to subject's treatment pathway plan post -procedure (discharge, surgeries such as bypass, amputation etc.) will be collected to determine patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

* Has symptomatic non-acute limb ischemia, requiring treatment of an infrainguinal artery
* Has Rutherford Clinical Category of 2-6
* is able and willing to provide written informed consent prior to study procedure

Angiographic Inclusion Criteria

* 100% stenosis by a visual estimate of angiography at the time of the procedure
* target CTO has moderate to severe calcification
* Has at least one of the following: severe calcification, flush occlusion, femoropopliteal CTOs with reconstitution below Popliteal 2-3, side directing collateral at the proximal cap, long (≥ 5cm) occlusions, below the knee (BTK) occlusion.
* Has evidence of a clinically significant CTO located in a peripheral vessel below the infrainguinal ligament confirmed by angiography at time of the procedure.

Exclusion Criteria:

General Exclusion Criteria

* Insufficient kidney function or renal failure
* Subject has positive pregnancy test result
* Participation in any study of a study device, medication, biologic, or other agent during study or within 30 days prior to enrollment that is either a cardiovascular study or could, in the judgment of the investigator, affect the results of this study
* Subject in whom antiplatelet, anticoagulant therapy is contraindicated
* Uncorrectable bleeding diathesis, platelet dysfunction, thrombocytopenia with platelet count less than 100,000/ml or known coagulopathy
* Known, untreated allergy to contrast agents or medications used during or subsequent to endovascular intervention. Patients with aspirin allergy that have been desensitized are not excluded.
* History of heparin-induced thrombocytopenia (HIT) that cannot be treated with direct thrombin inhibitors.
* Psychiatric disorder which in the judgment of the investigator could interfere with provision of informed consent, completion of tests, therapy or general study compliance.

Angiographic Exclusion Criteria

* The target CTO is located < 3 cm from a stented segment.
* Has an acute or sub-acute intraluminal thrombus within the target vessel.
* Clinical/ angiographic evidence of distal embolization in the index extremity unresolved prior to crossing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-30 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Successful CTO Crossing assessed by angiographic imaging | at time of procedure
  Successful CTO Crossing using the SoundBite™ Crossing System (SCS)

SECONDARY OUTCOMES:
Successful luminal CTO crossing using the SCS with or without imaging assistance. | at time of procedure
  Luminal crossing defined as ≥50% true lumen passage as assessed by an independent imaging core lab.
Costs benefits associated with the use of the SCS compared to a retrospective randomly selected chart review of conventional PTA wire escalation at the clinical site. | through study completion; 15 months
  Imaging costs are excluded
Freedom from SCS related Major Adverse Events (MAE) at the time of procedure/discharge | at procedure until discharge; up to 48 hours
  MAEs examples: unplanned, index limb amputation, dissection of grade C or greater that require an intervention to resolve

CONTACTS AND LOCATIONS:
Overall Officials: George Adams, MD, Principal Investigator — Rex Hospital
Locations (2):
- Medical University of Graz, Graz, Austria
- Klinikum Hochsauerland GmbH, Klinik für Angiologie, Arnsberg, Germany

IPD SHARING:
Plan to Share IPD: No